CLINICAL TRIAL: NCT02933099
Title: Aprepitant for the Prevention of Chemotherapy-induced Nausea and Vomiting Following High-dose Cisplatin in Nasopharyngeal Carcinoma Patients：a Randomized Phase 3 Trial
Brief Title: Aprepitant for the Prevention of Chemotherapy-induced Nausea and Vomiting
Acronym: CINV
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ting Hu, MD, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: WuhanUHC
Record Dates: First submitted 2016-10-07; First posted 2016-10-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aprepitant arm (Experimental): Aprepitant+palonosetron+dexamethasone
  Interventions: Drug: Aprepitant+palonosetron+dexamethasone
- Control arm (Active Comparator): palonosetron+dexamethasone
  Interventions: Drug: palonosetron+dexamethasone

INTERVENTIONS:
Drug: Aprepitant+palonosetron+dexamethasone — Patients will receive the chemotherapy drugs as well as the following antiemetic drugs: aprepitant (125 mg orally on day 1 and 80 mg orally on days 2 and 3) plus palonosetron 0.25 mg IV and dexamethasone (20 mg orally on day 1 and 8 mg orally on days 2 and 3)
  Other Names: PDA
  Arms: Aprepitant arm
Drug: palonosetron+dexamethasone — Patients will receive the chemotherapy drugs as well as the following antiemetic drugs: palonosetron 0.25 mg IV and dexamethasone (12 mg orally on day 1 and 8 mg orally on days 2 and 3)
  Other Names: PD
  Arms: Control arm

SUMMARY:
To compare the antiemetic combination of palonosetron, dexamethasone, and aprepitant (PDA) with antiemetic combination of palonosetron and dexamethasone (PD) in nasopharyngeal carcinoma patients receiving docetaxel, cisplatin, and 5-FU based chemotherapy.

DETAILED DESCRIPTION:
Eligible patients will be randomized to receive different antiemetic regimens . In the experimental group,patients will receive aprepitant, palonosetron and dexamethasone .In the other group,patients will accept the same dose of palonosetron and dexamethasone. During the treatment, any grade of nausea and vomiting should be recorded in order to evaluate the complete response rate of CINV,nausea patients will be measured by a visual analogue scale (VAS) ,other adverse events should be recorded as well.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Histologically or cytologically confirmed nasopharyngeal carcinoma
3. Accept chemotherapy for the first time
4. Patients who will receive chemotherapy (docetaxel 60 mg/m2 intravenously (IV), cisplatin 60 mg/m2 IV, and 5-FU (5-Fluorouracil) 600 mg/m2 IV)
5. Written informed consent

Exclusion Criteria:

1. regnant or breast-feeding
2. Uncontrolled psychosis history
3. Inability or unwillingness to understand or cooperate with study procedures
4. Central nervous system tumors primary or secondary
5. Concurrent abdominal radiotherapy
6. History of uncontrolled diabetes mellitus
7. Patients of prostatic hyperplasia ，paralytic ileus，narrow feet glaucoma.
8. Known cardiac arrhythmia, uncontrolled congestive heart failure ,or acute myocardial infarction with the previous six month
9. Pre-existing nausea or vomiting
10. Inadequate hematological function and abnormal liver and renal function.
11. History of sensitivity to olanzapine
12. Concurrent application of quinolone antibiotic therapy
13. Treatment with another antipsychotic agent such as risperidone,quetiapine, clozapine,phenothiazine,or butyrophenone for 30 days prior to or during the chemotherapy.
14. Cytochrome P450 3A4 substrates within 7 days (terfenadine, cisapride, astemizole, pimozide)
15. Concurrent application of systemic corticosteroids
16. Active infection or gastrointestinal dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-04 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Complete response | Up to 10 days
  The primary endpoint is the rate of patients achieving a complete response(defined as no emetic episode and no use of rescue medication) during over all time (0 to 120 hours post chemotherapy)

SECONDARY OUTCOMES:
Acute Phase Response | 0 to 24 hours post chemotherapy
  To determine the effect on complete response(defined as no emetic episode and no use of rescue medication) rates in the acute (0 to 24 hours) phase of CINV.
Delayed Phase Response | >24 to 10 days post chemotherapy
  To determine the effect on complete response (defined as no emetic episode and no use of rescue medication)rates in the delayed (>24 to 120 hours post chemotherapy) phase of CINV.
Functional Living Index -Emesis (FLIE) | Up to 10 days
Safety and tolerability as measured by the incidence and severity of adverse | Up to 10 days
  To evaluate the safety and tolerability by the incidence and severity of adverse events during the treatment (0 to 120 hours post chemotherapy)

IPD SHARING:
Plan to Share IPD: Undecided